CLINICAL TRIAL: NCT05537298
Title: Cellular and Physical Function Outcomes Leading to Failed Muscle Recovery After Critical Illness
Brief Title: Muscle Recovery After Critical Illness
Acronym: TRACER
Status: Recruiting | Type: Observational
Sponsor: Kirby Mayer (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Oklahoma Medical Research Foundation (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Kirby Mayer, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 77407; 5K23AR079583 (NIH); R01AR081002 (NIH)
Record Dates: First submitted 2022-07-27; First posted 2022-09-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: ICU Acquired Weakness; Post Intensive Care Unit Syndrome; Muscle Weakness; Critical Illness
Keywords: skeletal muscle; physical function
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and muscle tissue will be collected from a subset of individuals (n = 32) at three time-points in recovery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivor: Patients (n = 209) surviving critical illness will be enrolled to longitudinal, observational study examining muscle strength, power, and fatigue as well as physical function at hospital discharge and repeated at 3-, 6-, and 12-month following. A subset of individuals (n =32) will undergo muscle biopsies and blood will be collected.
- Control: A group of healthy controls will be recruited to serve as comparator to measures of strength, power, physical function, and muscle tissue analyses. Controls will participate in a one-time assessment.

SUMMARY:
The overarching goal of the proposed study is to determine the trajectories of physical recovery and cellular markers involved with the underlying failure to recover muscle after critical illness, while exploring which characteristics are associated with sustained physical disability. This proposal will examine muscle pathophysiology carefully aligned with physical function outcomes in order to longitudinally assess the recovery, or failed recovery, of muscle function in participants after critical illness:

1. to examine the recovery of muscle and physical function in ICU survivors through longitudinal assessments
2. to investigate the underlying cellular markers and mechanisms of muscle recovery in ICU survivors
3. to determine which cellular markers contribute to physical disability in ICU survivors up to 1 year after hospital admission

DETAILED DESCRIPTION:
Patients surviving critical illness develop significant impairments in skeletal muscle, commonly referred to as ICU-acquired weakness (ICUAW)[8-10]. It is estimated that up to 70-80% of patients admitted to ICU will develop some degree of neuromuscular dysfunction, weakness, myopathy or atrophy [11,12]. ICUAW encompasses muscle impairments that develop as a direct result of admission for critical illness[13] and is an independent predictor of mortality and long-term functional impairments[14-19]. Interventions to mitigate muscle deficits and improve physical function are a critical area of rehabilitation because of the high prevalence of short- and long-term impairments. ICU survivorship is particularly important as roughly 6 million Americans will survive an acute admission to the ICU this year alone.[24-26] Survivors of critical illnesses such as sepsis, viral-illnesses including coronaviruses, and acute respiratory failure (ARF) have reduced quality of life, lost wages from inability to return to work and increased caregiver and healthcare burden for years after hospital discharge.[27-31] Impairments in skeletal muscle are known contributors to physical disability and specifically prevent the performance of simple daily life activities like standing up from a chair. However, very little is known about cellular mechanisms leading to muscle and physical dysfunction in patients surviving critical illness during recovery. These gaps in knowledge are significant because identifying the phenotypes and underlying cellular mechanisms that lead to impaired muscle and physical function will facilitate the development of pharmacologic and non-pharmacologic interventions to mitigate or reverse disability. From a scientific perspective, this proposal is noteworthy because it will be the first to assess muscle protein synthesis rates in combination with cellular phenotypes, muscle strength, and physical function in patients recovering from an ICU admission. Studying muscle at the cellular level and integrating that knowledge with physical function will help improve our understanding of why certain patients fail to recover.

Elucidating cellular mechanisms during recovery phase will provide the framework to develop interventions in subsequent studies. We will assess measures of muscle and physical function in the first year of recovery to establish why some patients have restored function, yet others have sustained disability. Improved classification of muscle dysfunction and physical function enables future studies to employ a targeted approach instead of the historical rehabilitation approach of one-size-fits-all. Specifically, the cellular findings will lead to development of novel interventions specifically designed for the underlying mechanisms, while identification of the recovery trajectories will enhance clinicians' ability to implement interventions to patients with the greatest need.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 y/o)
* admission for sepsis or acute respiratory failure with at least 72 hour stay in ICU

Exclusion Criteria:

* acute or chronic neurologic condition
* acute or chronic orthopedic condition preventing strength/functional testing
* patients who were not ambulatory prior to ICU admission
* patients not expected to survive ~6months after admission

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU for critical illness and expected to survive
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical function | the change from baseline to 12-months
  Short Physical Performance Battery
Mitochondrial function | the change from baseline to 12-months
  muscle mitochondrial respirometry
Muscle power | the change from baseline to 12-months
  lower-extremity muscle power (unilateral leg-press to record Watts)

SECONDARY OUTCOMES:
Physical activity | the change from baseline to 12-months
  actigraphy measuring steps per day
Functional mobility | the change from baseline to 12-months
  timed-up and go test
Cardiopulmonary endurance / exercise capacity | the change from baseline to 12-months
  6-minute walk test
self-reported health-related quality of life | the change from baseline to 12-months
  EuroQol-5Domains (EQ-5D) visual analog scale is a self-report of quality of life (0-100) with higher scores indicating a better perception of quality of life
Muscle strength | the change from baseline to 12-months
  lower-extremity muscle strength measured by hand-held dynamometry (kilogram of force)
Muscle morphology #1 | the change from baseline to 12-months
  myofiber size
Muscle morphology #2 | the change from baseline to 12-months
  myofiber type

CONTACTS AND LOCATIONS:
Overall Officials: Kirby P Mayer, PhD, Study Director — University of Kentucky
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Kentucky, Lexington, Kentucky
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Seguel F, Summers LA, Fresenko LE, Long DE, Scott LN, Slone SA, Shankara Bhaktula S, Wen Y, Miller BF, Morris PE, Salyer AL, Kalema AG, Montgomery-Yates AA, Dupont-Versteegden EE, Mayer KP; TRACER study group Collaborators. Trajectories of Recovery after ACutE and cRitical illness (TRACER): a prospective observational study protocol. BMJ Open. 2025 Nov 19;15(11):e108885. doi: 10.1136/bmjopen-2025-108885. PMID 41263932